CLINICAL TRIAL: NCT00400855
Title: A Randomised, Double-blind, Placebo-controlled, Incomplete Block, 4-period Crossover, Study to Investigate the Effects of 5-day Repeat Inhaled Doses of Fluticasone Propionate (BID, 50-2000 mcg) on Airway Responsiveness to Adenosine 5-monophosphate (AMP) Challenge When Delivered After the Last Dose in Mild Asthmatic Subjects.
Brief Title: Study on the Effects of an AMP Challenge on Asthmatic Patients Following Treatment With Fluticasone Propionate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SIG103337
Record Dates: First submitted 2006-11-15; First posted 2006-11-17 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
Keywords: Asthma; AMP challenge
MeSH Terms: conditions — Asthma | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- Arm 1 (Experimental): study drug
  Interventions: Drug: Fluticasone propionate

INTERVENTIONS:
Drug: Fluticasone propionate — Study drug

SUMMARY:
Inhaling AMP causes an inflammatory response in the lung. This study will investigate whether 5-days of treatment with fluticasone propionate protects the lung from responding to the AMP in this way.

DETAILED DESCRIPTION:
A randomised, double-blind, placebo-controlled, incomplete block, 4-period crossover study to investigate the effects of 5-day repeat inhaled doses of fluticasone propionate (BID, 50-2000 mcg) on airway responsiveness to adenosine-5'-monophosphate (AMP) challenge when delivered after the last dose in mild asthmatic subjects

ELIGIBILITY:
Inclusion Criteria:

* Female of non-childbearing potential
* Using appropriate contraception.
* Mild asthmatic, non (or ex) smokers.
* Has inflammatory response to AMP.
* Otherwise healthy, not using any steroids.

Exclusion Criteria:

* Have a history of life-threatening asthma, defined as an asthma episode, which required intubation and/or was associated with either hypercapnea, respiratory arrest or hypoxia seizures.
* Have a known sensitivity to corticosteroids.
* Have a history of milk protein allergy.
* Test positive at the screening visit for hepatitis B or C or HIV

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2005-01; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
To characterise the dose response curve following repeat inhaled doses of FP for 5 days in the AMP challenge model. | 5 days

SECONDARY OUTCOMES:
Safety following multiple AMP challenges: Adverse events | 5 days
Plasma concentrations of FP and derived pharmacokinetic parameters | 5 days
Exhaled nitric oxide concentrations | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- New Zealand (2):
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Wellington

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: SIG103337 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: SIG103337 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SIG103337 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: SIG103337 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: SIG103337 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: SIG103337 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: SIG103337 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register